CLINICAL TRIAL: NCT03965403
Title: Upper Extremity Rehabilitation With the BURT Robotic Arm: a Feasibility Study
Brief Title: Upper Extremity Rehabilitation With the BURT Robotic Arm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Principal Investigator, Director of the Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016P002590
Record Dates: First submitted 2019-04-03; First posted 2019-05-29 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke; hemiparesis; Robotic
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm motor function retraining with BURT (Experimental): All participants will receive 1 hour sessions, 2-3x/week for 6 weeks (total 18 sessions). Sessions will be organized with 30 minutes of robotic-assisted training and 30 minutes of hands-on training with a research therapist to work on the baseline goals of the subject. Hands-on training will be done with routinely employed techniques in therapy to transfer the skills gained with the robotic device in everyday life activities.
  Interventions: Device: Arm motor function retraining with BURT

INTERVENTIONS:
Device: Arm motor function retraining with BURT — Intervention will be focused on patients impairments to assess the feasibility of the BURT device to carry-on long interventions

SUMMARY:
The overall objective of the proposed study is to carry out usability and design-evaluation assessments of the BURT robotic device for delivering long-term intervention in stroke survivors. The BURT is an upper extremity robotic device that enables the user to see and feel engaging games that encourage intensive therapy. The investigators intend to recruit up to 10 stroke survivors over the course of the study. Participants will train their arm with the BURT for 18 sessions over approximately 6 weeks then participate in a question/answer formatted discussion with research staff to discuss the usability of the device. The investigators will also assess participant's arm function at baseline and after the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age 18-80;
* Having had a stroke (ischemic or hemorrhagic) at least 6 months prior to study
* Moderate to severe upper-limb motor impairments (score of 15-45 out of 66 on the Fugl- Meyer Scale);
* Community dwelling;
* Able to physically fit in the device.

Exclusion Criteria:

* Current participation in rehabilitation program targeting upper extremity function;
* Cognitive impairment resulting to inability to follow instructions or inability to sustain attention for more than 10 minutes;
* Visual impairments not corrected with lenses (visual loss);
* Aphasia sufficient to limit comprehension and completion of the treatment protocol;
* No more than moderate impairments in paretic UE sensation, passive range of motion, and pain that would limit ability to engage in therapy;
* Increased muscle tone (passive movement is difficult);
* Previous diagnosis of neurological diseases other than stroke;
* Other conditions affecting function of the stroke affected upper limb;
* Individuals who present with the following: open wounds, fragile skin, active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm Motor Function Retraining With BURT
Started | 7
Completed | 6
Not Completed | 1
Not completed — Subject not meeting eligibility criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.38 (3.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Fugl-Meyer Upper Extremity Scores
Description: Assessment of upper extremity impairments. Individual items of the scale are summed for a total score ranking from 0 to 66. Higher scores indicate better outcomes.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 6
score on a scale | 3.50 (5.79)

2. Secondary Outcome: Changes From Baseline in Goal Attainment Scale Scores
Description: Standardized measure of goals selection and scaling to calculate the extend to which the participant's goals are met.
  The Goal Attainment Scale ranges from -2 to +2. Positive scores indicates goals are better than expected, score of 0 indicates goals are met and negative scores indicates goals aren't met.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 6
score on a scale | 0.22 (0.65)

3. Other Pre Specified Outcome: Changes From Baseline in Wolf Motor Function Test Scores (Time Subscale)
Description: Assessment of upper-extremity function by the performance time of the Wolf Motor Function Test). The average of the 15 items is reported. The time ranges from 0 to 120 seconds. A decrease in performance time is associated with improved upper-extremity function.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Time (seconds)
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 6
Time (seconds) | -6.43 (11.30)

4. Other Pre Specified Outcome: Changes From Baseline in Motor Activity Log Scores
Description: Use of upper extremity in daily life. The self-reported amount of use is reported on a scale from 0 to 5. A score of zero is assigned when the hemiparetic side is not used during the activity of daily living, a score of 5 is assigned when the hemiparetic side is used as much as before the stroke. The 30 items of the scale are averaged. Higher scores are a sign of better use in daily life.
Time Frame: 6 weeks
Population: One study participant did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 5
score on a scale | 0.42 (0.46)

5. Other Pre Specified Outcome: Changes From Baseline in Modified Ashworth Scale Scores
Description: Assessment of muscle tone for upper extremity muscles. Score rank from 0 (no tone) to 4 (no movement possible). Lower scores indicates a better outcome.
  Tone at the shoulder and elbow were measured
Time Frame: 6 weeks
Population: One study participant did not completed this evaluation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 5
score on a scale
  Shouder flexors | -0.1 (0.5)
  Shoulder extensors | 0.1 (0.9)
  Elbow flexors | 0.3 (0.7)
  Elbow extensors | 0.1 (1.1)
  Wrist flexors | -0.6 (0.8)
  Wrist extensors | -0.2 (0.8)
  Finger flexors | -0.5 (0.5)
  Finger extensors | 0.0 (0.0)

6. Other Pre Specified Outcome: Changes From Baseline in Articulations Range of Motion
Description: Assessment of active arm range of motion with goniometry. Results are reported in degrees and higher ranges include better outcomes.
Time Frame: 6 weeks
Population: One study participant did not complete this evaluation
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 5
degrees
  Shoulder Flexion | 5.00 (10.61)
  Shoulder extension | 14.6 (9.8)
  Shoulder ABD | 5.4 (10.9)
  Shoulder ADD | 3.4 (15.6)
  Shoulder IR | 0 (0)
  Shoulder ER | -5 (10)
  Elbow Flexion | 7.0 (10.4)
  Elbow extension | 1.0 (27.7)
  Forearm pronation | 2.0 (10.9)
  Forearm supination | 7.0 (12.0)
  Wrist extension | -2.0 (9.1)
  Wrist flexion | 14.0 (12.9)
  Ulnar flexion | 5.6 (5.2)
  Radial flexion | 1.0 (10.8)
  Index flexion | 9.0 (20.1)
  Index extension | -5.0 (8.7)

7. Other Pre Specified Outcome: Changes From Baseline in Manual Muscle Testing Scale Scores
Description: Assessment of arm muscle strength using the manual muscle testing scale ranking from 0 (no contraction) to 10 (maximal strength). Higher scores indicate better outcomes.
Time Frame: 6 weeks
Population: One study participant did not completed this evaluation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 5
score on a scale
  Shoulder flexors | 0.8 (1.1)
  Shoulder extensors | 1.6 (1.1)
  Shoulder adductors | 1.5 (1.6)
  Shoulder abductors | -0.2 (1.9)
  Shoulder internal rotators | 0.2 (1.1)
  Shoulder external rotators | 0.3 (1.1)
  Elbow flexors | 1.4 (1.1)
  Elbow extensors | 0.8 (3.6)
  Forearm pronators | 1.4 (3.6)
  Forearm supinators | -0.3 (1.6)
  Wrist extension | 0.1 (2.6)
  Wrist flexion | 1.5 (3.7)

8. Other Pre Specified Outcome: Changes From Baseline in Wolf Motor Function Test Scores (FAS Subcale)
Description: Assessment of upper-extremity function with the Functional ability subscale of the Wolf Motor Function Test.
  The average of the 15 items is reported. Scores ranges from 0 to 5, they rate the quality of the movement performance. 0= do not attempt, up to 5= identical to contralateral side. Higher scores are associated with better movement quality.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Motor Function Retraining With BURT
Number analyzed (Participants) | 6
score on a scale | 0.26 (0.37)

ADVERSE EVENTS:
Time Frame: We collected information in regard to potential adverse events during the 6 weeks of the study intervention.
Arm/Group | Arm Motor Function Retraining With BURT
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT03965403/Prot_000.pdf